CLINICAL TRIAL: NCT03795922
Title: A Multicenter, Double-blind, Randomized, Placebo-controlled, Parallel-group Study to Evaluate the Safety and Efficacy of MT10109L (NivobotulinumtoxinA) for the Treatment of Glabellar Lines
Brief Title: MT10109L in the Treatment of Glabellar Lines
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medy-Tox (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MT10109L-001; 2018-004384-31 (EudraCT Number)
Record Dates: First submitted 2018-12-20; First posted 2019-01-08 (Actual); Results first posted 2023-06-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Glabellar Lines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MT10109L (Experimental): MT10109L will be injected into the GL: initial double-blind treatment on Day 1, and up to 2 open-label study interventions during the retreatment period.
  Interventions: Drug: MT10109L
- Placebo (Placebo Comparator): Placebo will be injected into the GL: initial double-blind treatment on Day 1.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MT10109L — MT10109L will be injected into the GL.
  Other Names: NivobotulinumtoxinA
  Arms: MT10109L
Drug: Placebo — Placebo will be injected into the GL.
  Arms: Placebo

SUMMARY:
To evaluate the safety and efficacy of MT10109L in the treatment of glabellar lines (GL) in participants with moderate to severe GL.

ELIGIBILITY:
Inclusion Criteria

• Female participants must not be pregnant or planning to get pregnant and willing to minimize the risk of inducing pregnancy for the duration of the clinical study and follow-up period.

Exclusion Criteria

* Known immunization or hypersensitivity to any botulinum toxin serotype.
* Any medical condition that may put the participant at increased risk with exposure to MT10109L including diagnosed myasthenia gravis, Eaton Lambert syndrome, amyotrophic lateral sclerosis, or any other condition that might interfere with neuromuscular function.
* History of facial nerve palsy.
* Any uncontrolled systemic disease.
* Anticipated need for treatment with botulinum toxin of any serotype for any reason during the study (other than study intervention).
* Anticipated need for surgery or overnight hospitalization during the study.
* Prior exposure to botulinum toxin of any serotype for any reason.
* Prior periorbital surgery, facial lift (full face or mid-face), thread lift, brow lift, or related procedures (eg, eyelid [blepharoplasty] and/or eyebrow surgery).
* Prior facial treatment with permanent soft tissue fillers, synthetic implantation (eg, Gore-Tex®), and/or autologous fat transplantation.
* Current enrollment in an investigational drug or device study or participation in such a study within 30 days of entry into this study.
* Females who are pregnant, nursing, or planning a pregnancy during the study.
* Participants who plan for an extended absence away from the immediate area of the study site that would preclude them from returning for all protocol-specified study visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2018-12-24 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2021-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: SangMi Park, Study Director — Medytox Inc.
Locations (15):
- United States (9):
  - Investigate MD, Scottsdale, Arizona
  - Art of Skin MD, Solana Beach, California
  - Weinkle Dermatology, Bradenton, Florida
  - Etre, Cosmetic Dermatology and Laser Center, New Orleans, Louisiana
  - Dermatology and Laser Surgery Center of New York, New York, New York
  - SkinSearch of Rochester, Inc., Rochester, New York
  - M3 Wake Research, Inc., Raleigh, North Carolina
  - Aventiv Research, Inc., Dublin, Ohio
  - Westlake Dermatology & Cosmetic Surgery, Austin, Texas
- Belgium (4):
  - Centre de la Fontaine, Loverval, Hainaut
  - Medical Skin Care, Sint-Truiden, Limburg
  - Universitair Ziekenhuis Brussel, Brussels
  - CHU Liege, Liège
- Russia (2):
  - Kazan State Medical University, Kazan', Tatarstan Republic
  - Medical Centre Capital-Zdorovie, Moscow

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 234 met the inclusion/exclusion criteria and were randomized.
Groups:
- Placebo/MT10109L: Placebo was injected into the Glabellar Lines (GL): initial double-blind treatment on Day 1. In the open-label part, participants who met retreatment criteria were allowed up to 2 MT10109L treatments.
- MT10109L/MT10109L: MT10109L was injected into the Glabellar Lines (GL): initial double-blind treatment on Day 1, and up to 2 open-label study interventions during the retreatment period.
Period: Overall Study
Arm/Group | Placebo/MT10109L | MT10109L/MT10109L
Started | 80 | 154
Completed | 67 | 129
Not Completed | 13 | 25
Not completed — Adverse Event | 2 | 1
Not completed — Withdrawal by Subject | 5 | 13
Not completed — Lost to Follow-up | 2 | 3
Not completed — Pregnancy | 0 | 1
Not completed — Physician Decision | 1 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Other (Early termination, COVID, Family issue) | 3 | 4

BASELINE CHARACTERISTICS:
Population: 234 participants were included in the Intent To Treat (ITT) population (80 participants in the placebo group and 154 participants in the MT10109L group).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo/MT10109L | MT10109L/MT10109L | Total
Number analyzed (Participants) | 80 | 154 | 234
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 77 | 141 | 218
  >=65 years | 3 | 13 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.4 (11.57) | 47.3 (12.64) | 47.0 (12.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 140 | 216
  Male | 4 | 14 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 10 | 13
  Not Hispanic or Latino | 77 | 144 | 221
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 6 | 8
  White | 76 | 146 | 222
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Participants With a ≥ 2-grade Improvement From Baseline on the Facial Wrinkle Scale With Photonumeric Guide (FWS) According to INVESTIGATOR AND PARTICIPANT Assessments of Glabellar Lines (GL) Severity at Maximum Frown at Day 30
Description: The primary efficacy measure is a composite endpoint and a participant is considered responder only if both the investigator and participant independently report a ≥ 2-grade improvement at Day 30 of Double-Blind Period from baseline. Both participant and investigator used FWS to assess GL severity. FWS is 4-grade scale (0 to 3): 0=none and 3=severe.
  The primary endpoint is achieved and recorded as a count only when BOTH INVESTIGATOR AND PARTICIPANT assess the improvement in FWS from baseline to be ≥ 2-grade improvement. Therefore, the primary endpoint is the proportion/percentage of participants who meet the dual assessment threshold of ≥2-grade improvement from baseline.
Time Frame: Day 30
Population: All primary and secondary efficacy analyses endpoints were carried out using the Intent-To-Treat (ITT) analysis set, which was defined as all participants who were randomized. Multiple imputation method was used for missing variables in primary efficacy endpoint. Analyses of the secondary efficacy variables were performed using observed data.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo/MT10109L | MT10109L/MT10109L
Number analyzed (Participants) | 80 | 154
Participants | 0 | 71

2. Secondary Outcome: The Percentage of Responders for Investigator Assessments of Glabellar Lines (GL) Severity at Maximum Frown Using the Facial Wrinkle Scale (FWS)
Description: The Percentage of Responders for Investigator Assessments of Glabellar Lines (GL) Severity at Maximum Frown Using the Facial Wrinkle Scale (FWS), where a Responder was defined as Achieving a ≥2-grade Improvement from Baseline at Maximum Frown at Day 30 of double-blind period. The investigator evaluates the participant's GL severity using a 4-point scale (0 to 3) where 0=none and 3=severe
Time Frame: Day 30
Population: All secondary efficacy analyses were carried out using the Intent To Treat (ITT) analysis set, which was defined as all participants who were randomized. Analyses of the secondary efficacy variables were performed using observed data.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo/MT10109L | MT10109L/MT10109L
Number analyzed (Participants) | 77 | 153
Participants | 1 | 94

3. Secondary Outcome: The Duration of Glabellar Lines (GL) Treatment in Participants Who Achieved a Rating of ≥ 2-grade Improvement From Baseline in GL Severity at Maximum Frown at Day 30 According to Investigator Assessments Using the Facial Wrinkle Scale (FWS)
Description: The investigator evaluates the participant's GL severity using a 4-grade scale (0 to 3) where 0=none and 3 = severe. The outcome is measured as median time to loss of treatment effect (i.e., return to moderate or severe GL severity at maximum frown using the FWS).
Time Frame: Day 1 (first treatment) to Day 180
Population: The analysis population for this outcome includes the participants who achieved a rating of ≥ 2-gradeimprovement from baseline in GL severity at maximum frown at Day 30 of double-blind period according to investigator assessments using the Facial Wrinkle Scale (FWS). This corresponds to the responders for Outcome 2. Note: Analyses of the secondary efficacy variables were performed using observed data.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Placebo/MT10109L | MT10109L/MT10109L
Number analyzed (Participants) | 1 | 94
Days | 64 [NA to NA] — 95% Confidence Interval cannot be calculated as there was only 1 responder. | 121 [113 to 145]

4. Secondary Outcome: The Percentage of Participants Reporting Mostly Satisfied/Very Satisfied on the Facial Line Satisfaction Questionnaire (FLSQ) Follow-up Version Item 5 for Glabellar Lines (GL)
Description: The Satisfaction Question 5 grades facial line treatment satisfaction on a 5-point scale (-2 to 2) where -2=Very dissatisfied and 2=Very satisfied.
Time Frame: Day 60
Population: All secondary efficacy analyses were carried out using the Intent To Treat (ITT) analysis set, which wasdefined as all participants who were randomized. Analyses of the secondary efficacy variables wereperformed using observed data
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo/MT10109L | MT10109L/MT10109L
Number analyzed (Participants) | 72 | 145
Participants | 7 | 121

5. Secondary Outcome: The Percentage of Responders for Investigator Assessments of Glabellar Lines (GL) Severity at Rest Using the Facial Wrinkle Scale (FWS).
Description: The outcome was measured among participants who Were rated at least mild at rest at baseline, where a Responder was defined as achieving a ≥1-grade improvement from Baseline at Day 30 of double-blind period. The investigator evaluates the participant's GL severity using a 4-point scale (0 to 3) where 0=none and 3=severe.
Time Frame: Day 30
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo/MT10109L | MT10109L/MT10109L
Number analyzed (Participants) | 73 | 140
Participants | 23 | 95

6. Secondary Outcome: Number of Patients Who Experienced an Adverse Event (AE) Through the Study Duration
Description: This section focuses primarily on Treatment Emergent Adverse Events (TEAEs), i.e., AEs that started or worsened after the first dose of study intervention (Day 1) until up to 30 days after their last visit or study exit. The safety analyses were conducted in the Safety population. Unless otherwise noted, safety results refer to TEAEs.
Time Frame: The time frame for AEs is from the first dose on Day 1 and up to 30 days after their last visit or study exit (Day 360 or early exit).
Population: All safety analyses were carried out using the Safety population, defined as participants who received at least 1 dose of study intervention. Placebo participants who entered open-label phase (post Day 180) and received study intervention (MT10109L) are counted in MT10109L Group. Thus, overall number of participants in MT10109L Group is greater than what is noted in participant flow.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Placebo was injected into the Glabellar Lines (GL): initial double-blind treatment on Day 1. Placebo participants were allowed to enter open-label phase for retreatment but the TEAEs with onset date after the retreatment were not counted here.
- MT10109L: MT10109L was injected into the Glabellar Lines (GL): initial double-blind treatment on Day 1, and up to 2 open-label study interventions during the retreatment period. Placebo participants who experienced TEAE after receiving MT10109L during open-label phase were counted here.
Arm/Group | Placebo | MT10109L
Number analyzed (Participants) | 80 | 223
Participants | 35 | 118

7. Secondary Outcome: Mean Change From Baseline in Vital Signs - Systolic Blood Pressure (BP)
Description: Change from baseline at study exit.
Time Frame: Baseline to Study exit (Day 360 or early exit)
Population: All safety analyses were carried out using the Safety population subset at study exit , defined as participants who received at least 1 dose of study intervention. In order to calculate the mean change from baseline, participants with non-missing analysis values at both baseline and post-baseline during that analysis visit were used.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo/MT10109L | MT10109L/MT10109L
Number analyzed (Participants) | 73 | 133
mmHg | 0.3 (13.26) | -0.6 (15.28)

8. Secondary Outcome: Mean Change From Baseline in Vital Signs - Diastolic Blood Pressure (BP)
Description: Change from baseline at study exit.
Time Frame: Baseline to Study exit (Day 360 or early exit)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo/MT10109L | MT10109L/MT10109L
Number analyzed (Participants) | 73 | 133
mmHg | 0.5 (10.04) | -1.9 (10.64)

9. Secondary Outcome: Mean Change From Baseline in Vital Signs - Pulse Rate
Description: Change from baseline at study exit.
Time Frame: Baseline to Study exit (Day 360 or early exit)
Population: All safety analyses were carried out using the Safety population subset at study exit, defined as participants who received at least 1 dose of study intervention. In order to calculate the mean change from baseline, participants with non-missing analysis values at both baseline and post-baseline during that analysis visit were used.
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Placebo/MT10109L | MT10109L/MT10109L
Number analyzed (Participants) | 73 | 133
beats/min | 2.5 (10.35) | 0.4 (10.54)

10. Secondary Outcome: Mean Change From Baseline in Vital Signs - Respiratory Rate
Description: Change from baseline at study exit.
Time Frame: Baseline to Study exit (Day 360 or early exit)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: breaths/min
Arm/Group | Placebo/MT10109L | MT10109L/MT10109L
Number analyzed (Participants) | 73 | 133
breaths/min | -0.3 (2.44) | -0.3 (2.18)

11. Secondary Outcome: Mean Change From Baseline in Electrocardiogram (ECG) Parameters - Heart Rate
Description: Change from baseline at study exit.
Time Frame: Baseline to Study Exit (Day 360 or early exit)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Placebo/MT10109L | MT10109L/MT10109L
Number analyzed (Participants) | 70 | 130
beats/min | 4.8 (10.38) | 2.8 (8.52)

12. Secondary Outcome: Mean Change From Baseline in Electrocardiogram (ECG) Parameters - PR Interval
Description: Change from baseline at study exit.
Time Frame: Baseline to Study Exit (Day 360 or early exit)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo/MT10109L | MT10109L/MT10109L
Number analyzed (Participants) | 70 | 130
milliseconds | -1.2 (11.67) | -1.2 (11.91)

13. Secondary Outcome: Mean Change From Baseline in Electrocardiogram (ECG) Parameters - QRS Duration
Description: Change from baseline at study exit.
Time Frame: Baseline to Study Exit (Day 360 or early exit)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo/MT10109L | MT10109L/MT10109L
Number analyzed (Participants) | 70 | 130
milliseconds | 0.4 (6.65) | 1.2 (6.41)

14. Secondary Outcome: Mean Change From Baseline in Electrocardiogram (ECG) Parameters - QT Interval
Description: Change from baseline at study exit.
Time Frame: Baseline to Study Exit (Day 360 or early exit)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo/MT10109L | MT10109L/MT10109L
Number analyzed (Participants) | 70 | 130
milliseconds | -11.7 (23.87) | -8.4 (19.71)

15. Secondary Outcome: Mean Change From Baseline in Electrocardiogram (ECG) Parameters - QTcB Interval
Description: Change from baseline at study exit.
Time Frame: Baseline to Study Exit (Day 360 or early exit)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo/MT10109L | MT10109L/MT10109L
Number analyzed (Participants) | 70 | 130
milliseconds | 2.7 (18.69) | 0.0 (17.14)

16. Secondary Outcome: Mean Change From Baseline in Electrocardiogram (ECG) Parameters - QTcF Interval
Description: Change from baseline at study exit.
Time Frame: Baseline to Study Exit (Day 360 or early exit)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo/MT10109L | MT10109L/MT10109L
Number analyzed (Participants) | 70 | 130
milliseconds | -2.4 (15.43) | -2.9 (14.06)

17. Secondary Outcome: Mean Change From Baseline in Electrocardiogram (ECG) Parameters - RR Interval
Description: Change from baseline at study exit.
Time Frame: Baseline to Study Exit (Day 360 or early exit)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo/MT10109L | MT10109L/MT10109L
Number analyzed (Participants) | 70 | 130
milliseconds | -64.6 (127.1) | -39.3 (106.19)

18. Secondary Outcome: Number of Participants With Binding and Neutralizing Antibodies
Description: Only samples that tested positive in the binding antibody confirmatory assay were evaluated for neutralizing antibodies. The participants with positive neutralizing antibodies are only shown.
Time Frame: Up to Study Exit (Day 360 or early exit)
Population: All safety analyses were carried out using the Safety population subset at study exit , defined as participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo/MT10109L | MT10109L/MT10109L
Number analyzed (Participants) | 80 | 154
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: The time frame for AEs is from the first dose on Day 1 and up to 30 days after their last visit or study exit (Day 360 or early exit).
Description: All safety analyses were carried out using the Safety population, defined as participants who received at least 1 dose of study intervention. Placebo participants who entered open-label phase (post Day 180) and received study intervention (MT10109L) are counted in MT10109L Group. Thus, overall number of participants in MT10109L Group is greater than what is noted in participant flow.
Groups:
- Placebo: Placebo was injected into the Glabellar Lines (GL): initial double-blind treatment on Day 1. In the open-label part post day 180, up to 2 open-label study interventions during the retreatment period. Placebo participants were allowed to enter open-label phase for retreatment but the TEAEs with onset date after the retreatment were not counted here.
Arm/Group | Placebo | MT10109L
All-Cause Mortality (participants affected / at risk) | 0/80 | 0/223
Serious Adverse Events (participants affected / at risk) | 3/80 | 5/223
Other Adverse Events (participants affected / at risk) | 8/80 | 32/223
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=80) | MT10109L (N=223)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Rectal prolapse (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast Cancer Stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant Melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Intentional Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=80) | MT10109L (N=223)
Headache (Nervous system disorders) | 4 (4) | 22 (22)
Injection site pain (General disorders) | 4 (4) | 16 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
General research agreement between the sponsor and PI's that includes a confidentiality section that includes a statement that the sponsor is and shall remain the exclusive owner of 'Information'. 'Information' shall include, but shall not be limited to, protocols, trade secrets, know-how, formulations, inventions, techniques, equipment, data and results.

DOCUMENTS (2):
  • Study Protocol (2020-09-30): https://cdn.clinicaltrials.gov/large-docs/22/NCT03795922/Prot_002.pdf
  • Statistical Analysis Plan (2020-11-18): https://cdn.clinicaltrials.gov/large-docs/22/NCT03795922/SAP_003.pdf